CLINICAL TRIAL: NCT01044056
Title: An Open-label, Randomized, Parallel Group Trial in Healthy Female Subjects to Compare the Pharmacokinetics of Ethinyl Estradiol of NuvaRing®, a Contraceptive Patch (EVRA(TM)) and an Oral Contraceptive (Microgynon® 30)
Brief Title: A Trial in Healthy Female Subjects to Compare the Pharmacokinetics of Ethinyl Estradiol of NuvaRing®, a Contraceptive Patch (EVRA(TM)) and an Oral Contraceptive (Microgynon® 30) (Study 34237 (P06650)) (COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P06650
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception
MeSH Terms: interventions — Levonorgestrel; Contraceptives, Oral; ethinyl estradiol, levonorgestrel drug combination; Ortho Evra; NuvaRing; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Levonorgestrel/ethinylestradiol oral contraceptive pill (Active Comparator): Microgynon(R), 1 tablet every day for 21 days; each tablet contains 0.150 mg levonorgestrel (LNG) and 0.030 mg ethinylestradiol (EE).
  Interventions: Drug: Levonorgestrel (LNG)/Ethinylestradiol (EE) oral contraceptive tablets
- Norelgestrominum and ethinylestradiol contraceptive patch (Active Comparator): Evra(TM), One patch applied on lower abdomen for 7 days for 3 consecutive weeks, 3 patches in total. Each patch contains 6 mg norelgestromin and 0.750 mg EE releasing 0.150 mg norelgestromin and 0.020 mg EE per day.
  Interventions: Drug: norelgestrominum and ethinylestradiol patch oral contraceptive patch
- Etonogestrel and ethinylestradiol contraceptive vaginal ring (Active Comparator): Nuvaring(R), Place the ring in the vagina for 21 days, remove for one week. Repeat with new Ring. Dose: per ring 11.7 mg ENG and 2.7 mg EE releasing a daily average amount of 0.120 mg ENG and 0.015 mg EE.
  Interventions: Drug: Nuvaring ™ (etonorgestrel/ethinylestradiol)

INTERVENTIONS:
Drug: Levonorgestrel (LNG)/Ethinylestradiol (EE) oral contraceptive tablets — LNG/EE oral contraceptive tablets (Microgynon® 30), 21 in total, containing 0.150 mg LNG and 0.030 mg EE per tablet administered once daily orally for 21 consecutive days.
  Other Names: Microgynon; Batch Number: 374A 01K05
  Arms: Levonorgestrel/ethinylestradiol oral contraceptive pill
Drug: norelgestrominum and ethinylestradiol patch oral contraceptive patch — A contraceptive patch (EVRA ™), one patch for 7 days for three consecutive weeks, 3 patches in total, applied on the lower abdomen. Dose: per patch 6 mg norelgestromin and 0.750 mg EE releasing 0.150 mg norelgestromin and 0.020 mg EE per day.
  Other Names: EVRA ™; Batch number : 0311264
  Arms: Norelgestrominum and ethinylestradiol contraceptive patch
Drug: Nuvaring ™ (etonorgestrel/ethinylestradiol) — NuvaRing ™ , one ring for a period of 21 days, inserted vaginally. Dose: per ring 11.7 mg etonogestrel and 2.7 mg EE releasing a daily average amount of 0.120 mg etonogestrel and 0.015 mg EE.
  Arms: Etonogestrel and ethinylestradiol contraceptive vaginal ring

SUMMARY:
An open-label, randomized, parallel group trial in healthy female subjects to compare the pharmacokinetics of ethinyl estradiol (EE) of NuvaRing®, a contraceptive patch (EVRA(TM)) and an oral contraceptive (Microgynon® 30).

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 but not older than 40 years of age on Day 1 of treatment.
* Subject has uterus and ovaria in situ
* Subject who does not use hormonal contraception and is willing to use adequate nonhormonal contraceptive measures during the timeframe between screening and start treatment.
* Subject is able and willing to refrain from caffeine and/or xanthine containing food and/or beverages (e.g. coffee, tea, cola or chocolate) from 24 hours before the first administration of the trial medication until the last PK blood sample.
* Subject is willing not to consume grapefruit containing products 14 days prior to the start of the first administration of the trial medication until the last PK blood sample.
* Subject is willing to refrain from smoking from 7 days prior to first administration of the trial medication until the last pharmacokinetic blood sample.
* Subject is willing to refrain from alcohol containing products from 24 hours prior to first administration of the trial medication until the last pharmacokinetic blood sample.

Exclusion Criteria:

* Contraindications for use of NuvaRing, contraceptive patch and oral contraceptive:
* Presence or history of venous thrombosis, with or without the involvement of pulmonary embolism.
* Presence or history of arterial thrombosis (e.g. cerebrovascular accident, myocardial infarction) or prodromi of a thrombosis (e.g. angina pectoris or transient ischaemic attack).
* Known predisposition for venous or arterial thrombosis, with or without hereditary involvement such as Activated Protein C (APC) resistance, antithrombin-III deficiency, protein C deficiency, protein S deficiency, hyperhomocysteinaemia, antiphospholipid antibodies (anticardiolipin antibodies, lupus anticoagulant) and Factor V Leiden mutation.
* Diabetes mellitus with vascular involvement
* The presence of a severe or multiple risk factor(s) for venous or arterial thrombosis (to be judged by the (sub-) investigator
* Presence or history of severe hepatic disease as long as liver function values had not returned to normal or were judged to be clinically significant by the investigator.
* Presence or history of liver tumours (benign or malignant).
* Known or suspected malignant conditions of the genital organs or the breasts, if sex-steroid-influenced.
* Undiagnosed vaginal bleeding.
* Hypersensitivity to the active substances or to any of the excipients of NuvaRing, contraceptive patch and oral contraceptive.
* Migraine with focal aura
* Known or suspected pregnancy
* Breastfeeding, or within 2 months after stopping breastfeeding on the day preceding the first administration of trial medication (Day -1).
* Clinically significant abnormal laboratory, ECG (electrocardiogram) vital signs, physical and gynecological findings at screening.
* A significant (history of) allergic or other serious disease, particularly gastrointestinal tract disease.
* Smoking more than 5 cigarettes or 1 pipe or 1 cigar per day for a period of at least 3 months prior to screening.
* Using any systemic medication (including over the counter (OTC) medication) during the 14 days prior to the day preceding the first administration of trial medication (Day -1), except for oral contraceptive used for synchronization and occasional Ibuprofen.
* Used any drug or substance that is known to induce drug-metabolizing enzymes within two months prior to the start of synchronization.
* Received a contraceptive by injection, an implant or hormonal intra-uterine device within 6 months of the day preceding the first administration of trial medication (Day -1), or a hormonal implant or hormonal intra-uterine device removed within 6 months of the day preceding the first administration of trial medication (Day -1).
* Participated in a drug trial and was administered an investigational drug during the 90 days prior to start of synchronization.
* Donated blood during the 90 days prior to the day preceding the first administration of trial medication (Day -1).
* History (within the last 2 years) of excessive alcohol use, use of solvents or of drug abuse.
* Positive drug test at screening and/or admission (Day -1), or a positive alcohol test at admission (Day -1).
* Clinically significant abnormal cervical smear result (papaninecolaou (PAP) III or higher) at screening.
* Acute or chronic hepatitis B/C or human immune deficiency virus (HIV) 1&2 infection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

REFERENCES:
- [Result] van den Heuvel MW, van Bragt AJ, Alnabawy AK, Kaptein MC. Comparison of ethinylestradiol pharmacokinetics in three hormonal contraceptive formulations: the vaginal ring, the transdermal patch and an oral contraceptive. Contraception. 2005 Sep;72(3):168-74. doi: 10.1016/j.contraception.2005.03.005. PMID 16102549

RESULTS

PARTICIPANT FLOW:
Groups:
- Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill: Levonorgestrel (LNG)/ethinylestradiol (EE) oral contraceptive tablets (Microgynon® 30), 21 in total, containing 0.150 mg LNG and 0.030 mg EE per tablet administered once daily orally for 21 consecutive days.
- Norelgestrominum and Ethinylestradiol Contraceptive Patch: A contraceptive patch (EVRA(TM)), one patch for seven (7) days for three consecutive weeks, three (3) patches in total, applied on the lower abdomen. Dose: per patch 6 mg norelgestromin and 0.750 mg EE releasing 0.150 mg norelgestromin and 0.020 mg EE per day.
- Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring: NuvaRing®, one ring for a period of 21 days, inserted vaginally. Dose: per ring 11.7 mg etonogestrel (ENG) and 2.7 mg EE releasing a daily average amount of 0.120 mg etonogestrel and 0.015 mg EE.
Period: Overall Study
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (5.44) | 24.8 (6.59) | 23.1 (3.64) | 24.5 (5.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 8 | 24
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration (Cmax) (Pharmacokinentic Parameter (PK)) for All Subjects in the Pharmacokinetically Evaluable (ASPE) Group
Description: Cmax was measured using ethinylstradiol serum concentration at several time points during the 21 days of active treatment and the washout thereafter.
Time Frame: 21 days of active treatment and washout period thereafter
Population: Subjects who received at least one dose of medication
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring
Number analyzed (Participants) | 8 | 6 | 8
pg/ml | 168 (29.5) | 105 (12.4) | 37.1 (5.1)

2. Primary Outcome: Area Under the Curve (AUC) 0-21 Days (PK Parameter) Measured for the ASPE Group
Description: AUC 0-21 days was measured using ethinylestradiol serum concentration using a radio-immune assay at several time points during the 21 days of active treatment
Time Frame: 21 days
Population: Subjects who received at least one dose of medication.
Measure: Mean (Standard Deviation); unit: nh.h/mL
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring
Number analyzed (Participants) | 8 | 6 | 8
nh.h/mL | 21.9 (2.9) | 35.8 (5.5) | 10.6 (2.5)

3. Primary Outcome: AUC 0-tlast (PK Parameter) for the ASPE Group.
Description: AUC 0-tlast was measured using ethinylestradiol serum concentrations using a radio-immune assay at several time points during the 21 days of active treatment and the washout period thereafter.
Time Frame: 21 days of active treatment and washout period thereafter
Population: Subjects who received at least one dose of medication.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring
Number analyzed (Participants) | 8 | 6 | 8
ng.h/mL | 22.5 (2.9) | 37.5 (5.7) | 11.1 (2.7)

4. Primary Outcome: AUC 0-infinity (PK Parameter) for the ASPE Group.
Description: AUC 0-infinity was measured using ethinylestradiol serum concentration using a radio-immune assay at several time points during the 21 days of active treatment and the washout period thereafter. AUC 0-infinity was calculated as AUC 0-tlast extrapolated to infinity using the regression line from which t 1/2 was calculated.
Time Frame: 21 days of active treatment and the washout period thereafter
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Pill | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring
Number analyzed (Participants) | 8 | 6 | 8
ng.h/mL | 22.7 (2.8) | 37.7 (5.6) | 11.2 (2.7)

ADVERSE EVENTS:
Time Frame: 21 days
Groups:
- Levonorgestrel/Ethinylestradiol Oral Contraceptive Tablets: Levonorgestrel (LNG)/ethinylestradiol (EE) oral contraceptive tablets (Microgynon(R) 30), 21 in total, containing 0.150 mg LNG and 0.030 EE per tablet administered once daily orally for 21 consecutive days.
- Norelgestrominum and Ethinylestradiol Contraceptive Patch: A contraceptive patch (EVRA(TM), one patch for 7 days for three consecutive weeks, 3 patches in total, applied on the lower abdomen. Dose: per patch 6 mg norelgetromin and 0.750 mg EE releasing 0.150 mg norelegestromin and 0.020 mg EE per day.
- Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring: Nuvaring(R), one nring for a period of 21 days, inserted vaginally. Dose: per ring 11.7 mg etonrgestrel (ENG) and 2.7 mg EE releasing a daily average amount of 0.120 mg etonorgestrel and 0.015 mg EE
Arm/Group | Levonorgestrel/Ethinylestradiol Oral Contraceptive Tablets | Norelgestrominum and Ethinylestradiol Contraceptive Patch | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levonorgestrel/Ethinylestradiol Oral Contraceptive Tablets (N=8) | Norelgestrominum and Ethinylestradiol Contraceptive Patch (N=8) | Etonogestrel and Ethinylestradiol Contraceptive Vaginal Ring (N=8)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 4 (6) | 1 (2)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
LOOSE STOOLS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 3 (6) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
APPLICATION SITE DERMATITIS (General disorders) | 0 (0) | 1 (1) | 0 (0)
APPLICATION SITE IRRITATION (General disorders) | 0 (0) | 2 (2) | 0 (0)
APPLICATION SITE PRURITUS (General disorders) | 0 (0) | 3 (4) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 3 (3) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
VENIPUNCTURE SITE PAIN (General disorders) | 1 (1) | 1 (1) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 1 (2) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ANIMAL SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 5 (9) | 4 (10)
SYNCOPE VASOVAGAL (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
MOOD ALTERED (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
BREAST TENDERNESS (Reproductive system and breast disorders) | 0 (0) | 5 (7) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
GENITAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (4) | 1 (1)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No